CLINICAL TRIAL: NCT04904263
Title: Advisory Board on Cancer, Infertility and Pregnancy
Acronym: ABCIP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Gasthuisberg (Other)
Collaborators: Kom Op Tegen Kanker (Other); European Research Council (Other)
Responsible Party: Principal Investigator, Frederic Amant, Prof. dr. Amant, University Hospital, Gasthuisberg
Other Study IDs: ABCIP
Record Dates: First submitted 2021-05-22; First posted 2021-05-27 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Cancer in Pregnancy; Fertility Preservation; Cancer; Pregnancy
Keywords: Cancer in Pregnancy; Fertility preservation
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Advisory Board on Cancer, Infertility and Pregnancy provides a platform where physicians from all over the world can request recommendations regarding the medical care of pregnant women diagnosed with cancer or regarding fertility preservation. The platform will contain different national advisory boards, with their own coordinator and members, as well as an overarching international advisory board with an international coordinator and members from different national boards.

To investigate the impact of this platform, a year after its launch, data regarding the incoming requests will be extracted from the website, as well as all recommendation letters.

DETAILED DESCRIPTION:
The Advisory Board on Cancer, Infertility and Pregnancy (ABCIP)-platform will be a web-based platform where clinicians from all over the world can request advice from a group of experts on the field of Cancer and Pregnancy. The platform will contain different national advisory boards, with their own coordinator and members, as well as an overarching international advisory board with an international coordinator and members from different national boards.

Clinicians can fill in a format (attached) requesting for advice, using only pseudonymized patient data after agreeing a disclaimer:

All information filled in in the 'request advice' format needs to be regarded as anonymous or pseudonymous data. We recommend you to inform your patient and ask for approval when needed, based on the rules and regulations applicable in your country.

The filled out request will be sent to the specific national board of their own country, and if no national board is available, to the overarching international board.

. To investigate the impact of this platform, a year after its launch, data regarding the incoming requests will be extracted from the website, as well as all recommendation letters.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with a cancer diagnosis
* Women with a fertility related question after cancer diagnosis
* Postpartum cancer diagnosis
* Cancer treatment during pregnancy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Advice can be requested regarding all patients with cancer during pregnancy, questions regarding patients with a fertility wish after cancer diagnosis or questions regarding patients with a postpartum cancer diagnosis
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-05-22 (Estimated); Primary Completion 2024-05-22 (Estimated); Study Completion 2024-05-22 (Estimated)

PRIMARY OUTCOMES:
The impact of an international advisory board on cancer in pregnancy | 1 year
  To investigate the impact of this platform, a year after its launch, data regarding the incoming requests will be extracted from the website, as well as all recommendation letters. All requesting physicians will be asked to complete a survey including their experiences with the ABCIP, to what amount they followed the given recommendations and the outcomes of mother (and child)

CONTACTS AND LOCATIONS:
Overall Officials: Frederic Amant, MD,PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- UZ Gasthuisberg, Katholieke Universiteit Leuven, Leuven, Belgium

REFERENCES:
- See also: Link to the ABCIP platform — http://www.ab-cip.org